CLINICAL TRIAL: NCT05072795
Title: MUSC Specialized Center of Research Excellence (SCORE) on Sex Differences: Stress-Reactivity and Cannabis Use in Cannabis-Using Older Adults
Brief Title: Stress-Reactivity and Cannabis Use in Cannabis-Using Older Adults
Acronym: PUMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Andreana Benitez, Assistant Professor, Medical University of South Carolina
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 00111432; 3U54DA016511-19S1 (NIH)
Record Dates: First submitted 2021-09-24; First posted 2021-10-11 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Cannabis Use

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Induction (Experimental): Participants completed the Trier Social Stress Test (TSST)
  Interventions: Behavioral: Trier Social Stress Task (TSST)
- No intervention (No Intervention): Participants did not complete the Trier Social Stress Test (TSST).

INTERVENTIONS:
Behavioral: Trier Social Stress Task (TSST) — The TSST is a standardized psychological stress challenge which provokes a stress response in a laboratory setting. During the task, saliva samples will be collected for hormone testing along with physiological and subjective measures.
  Arms: Stress Induction

SUMMARY:
The goal of the study is to evaluate how cannabis use affects memory and thinking skills and response to stress in older adults. The study will also relate cannabis use to Alzheimer's Disease (AD) biomarkers (measurable substances in blood that indicate condition), and test whether sex and hormones play a role in these effects. The study is recruiting adults between the ages of 50 and 80 who use cannabis products on a regular basis. Study participation will last about two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80.
* Women must be >1 year post-menopausal.
* English as a first/primary language.
* Functional visual and auditory acuity (aided or unaided) to complete tests.
* Capacity to independently provide informed consent and function at an intellectual level sufficient to allow completion of all instruments.
* Currently meets DSM-5 criteria for CUD or uses cannabis at least 4 days per week
* Consent to abstain from alcohol and cannabis use for >12 hours prior to Study Visit (Day 0), and TSST (Day 8).
* Consent to abstain from all drugs other than cannabis or nicotine for the duration of the study.

Exclusion Criteria:

* Meet DSM-5 criteria for moderate or severe alcohol or substance use disorder (other than nicotine or cannabis) within the last 12 months.
* History of major neurocognitive disorder or developmental disorder per DSM-5.
* A Telephone Interview for Cognitive Status (TICS) score of less than or equal to 22.
* Significant or unstable medical condition/s that impact cognition as deemed by study investigators, such as active significant cardiac, cerebrovascular, neoplastic, infectious, or metabolic disease, or longstanding and intractable severe mental illness (e.g. schizophrenia spectrum disorder, bipolar disorder).
* Daily use of medications that adversely impact cognition in aging (i.e. anticholinergics and sedatives).
* Current suicidal or homicidal ideation/risk.
* Unable to complete/comply with procedures or pose threat to research staff.
* Standard MRI contraindications (e.g., implants, claustrophobia).
* Women who are pregnant, nursing, or of childbearing potential and not practicing and effective means of birth control.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreana Benitez, PhD, Principal Investigator — Medical University of South Carolina; Aimee Aimee McRae-Clark, PharmD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between Oct 2021 and May 2023 through community advertisements.
  The first participant was enrolled on 11/19/2021 and the last participant was enrolled on 5/18/2023.
Pre-assignment Details: There was one participant group (N=47). All participants completed cognitive testing on Day 0 and a stress intervention on Day 8.
  Cognition was assessed independently of the stress intervention and is the primary outcome. N=47 completed the cognition assessments, which we listed as the non-intervention group. Stress intervention was not a primary outcome and is not reported in results section. N=45 completed the Stress Induction and are listed below.
Period: Overall Study
Arm/Group | Stress Induction
Started | 47
Completed | 42
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Stress Induction
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.11 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 42
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Global Cognitive Ability (GCA)
Description: The primary outcome is the mean Global Cognitive Ability (GCA) z-score, which is a psychometrically robust, factor analytically-derived, demographically-normed index of global cognitive function. A Z-score of 0 represents the population mean with positive scores indicating a higher level of cognitive function and negative scores indicating a lower level of cognitive function than the mean. The investigator will test the hypothesis that women with CUD will have lower GCA scores than men.
Time Frame: Day 0
Population: Hypothesis was that women with CUD will have lower GCA scores than men.
Measure: Mean (Standard Deviation); unit: Standard score (Z-score)
Groups:
- Independent of Intervention: No intervention
Arm/Group | Independent of Intervention
Number analyzed (Participants) | 47
Standard score (Z-score)
  Male: number analyzed (Participants) | 26
  Male | -1.99 (1.31)
  Female: number analyzed (Participants) | 21
  Female | -0.82 (1.37)
Statistical Analysis 1: Comparison: Independent of Intervention; Test type: Other; p = 0.005, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Stress Induction
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT05072795/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT05072795/ICF_000.pdf